CLINICAL TRIAL: NCT06100627
Title: A Randomized, Open-Label, Parallel Group, Phase 1 Study to Assess the Pharmacodynamic Effect of AP301 on Urinary Phosphorus Excretion in Healthy Volunteers
Brief Title: A Pharmacodynamic Effect Study of AP301 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alebund Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Alebund Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP301-PD-01
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy Subjects
Keywords: Pharmacodynamic; safety; tolerability; AP301; Healthy subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2.10 g/day of AP301 (Experimental)
  Interventions: Drug: AP301
- 4.20 g/day of AP301 (Experimental)
  Interventions: Drug: AP301
- 6.30 g/day of AP301 (Experimental)
  Interventions: Drug: AP301
- 8.40 g.day of AP301 (Experimental)
  Interventions: Drug: AP301

INTERVENTIONS:
Drug: AP301 — Orally administered

SUMMARY:
This is a randomized, open-label, parallel-group, phase 1 study to evaluate the PD effect of AP301 capsule in healthy volunteers. The study is planned to have 4 treatment arms: Arm 1: 2.10 g/day; arm 2: 4.20 g/day; arm 3: 6.30 g/day; arm 4: 8.40 g/day.

DETAILED DESCRIPTION:
A total of 32 participants will participate in this study and the study consists of 3 periods such as screening period, hospitalization period and follow up period.

ELIGIBILITY:
Important Inclusion Criteria:

* Healthy male volunteers, 18-55 years of age
* Body mass index (BMI) 18-30 kg/m2 (exclusive) at screening.

Important Exclusion Criteria:

* Serum phosphorus is below 1.00 mmol/L at screening.
* History of significant gastrointestinal disease or disorder, major gastrointestinal surgeries, or cholecystectomy
* History or symptoms of any clinically significant kidney, liver, broncho-pulmonary, gastrointestinal, neurological, psychiatric, cardiovascular, endocrine/metabolic, hematological diseases, or cancer.
* History of specific allergies or allergic conditions or known allergies to the study drug as judged by the investigator, or any confirmed significant allergic reactions (urticaria or anaphylaxis) to any drug, or multiple drug allergies (non-active hay fever is acceptable). Allowing for childhood asthma, history of mild eczema that has had no flare ups for ≥5 years or is fully resolved.
* Known history of allergy to common food like milk or gluten, or lactose intolerance, or special diet habit for religious/life-style reasons, which might potentially jeopardize the participant's compliance of study diet.
* Any clinically significant concomitant disease, or condition or treatment that could interfere with the conduct of the study.
* Confirmed (based on the average of 3 separate resting blood pressure measurements, after at least 5 minutes rest) systolic blood pressure (BP) greater than 150 or less than 90 mmHg, and diastolic BP greater than 90 or less than 50 mmHg at screening.
* Clinically relevant ECG abnormalities on screening ECG.
* Estimated glomerular filtration rate (eGFR) ≤ 70 mL/min/1.73 m2.
* Positive test at screening of any of the following: Hepatitis B (HBsAg), Hepatitis C (HCV Ab) or human immunodeficiency virus (HIV-1 or HIV-2 Ab).
* Alanine aminotransferase (ALT) or aspartate transaminase (AST) > 1.5 × upper limit of normal (ULN), or any other clinically significant abnormalities in laboratory test results at screening.
* Dosed with a small-molecule or biologic investigational drug within 30 days or 90 days, respectively, or 5 half-lives (whichever is the longer) prior to first dose of this study.
* Positive urine test for drugs of abuse and/or positive alcohol test at screening.
* Any medical or social conditions that, in the view of investigator, might potentially jeopardize the participant's compliance of study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 32 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Urinary phosphorus excretion during AP301 administration | From the Day 1 to Day 4 after dosing, assessed up to 3 days
  Average daily urinary phosphorus excretion during the 3 consecutive days of AP301 treatment
Effect of AP301 on urinary phosphorus excretion | From Day -3 to Day 4 after dosing, assessed up to 6 days
  Change of average daily urinary phosphorus excretion from 3 days before treatment to 3 days during treatment.
Urinary calcium excretion during AP301 administration | From the Day 1 to Day 4 after dosing, assessed up to 3 days
  Average daily urinary calcium excretion during the 3 consecutive days of AP301 treatment.
Effect of AP301 on urinary calcium excretion | From Day -3 to Day 4 after dosing, assessed up to 6 days
  Change of average daily urinary calcium excretion from 3 days before treatment to 3 days during treatment.
Effect of AP301 on serum phosphorus and calcium | From Day -3 to Day 4 after dosing, assessed up to 6 days
  Changes of serum phosphorus and serum calcium from baseline to end of treatment.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From screening to hospitalization and follow up periods, assessed up to 43 days
  Number of participants with adverse events (AEs) and the intensity of adverse events.
  Number of participants with serious adverse events (SAEs) and the intensity of adverse events.
Changes in clinical laboratory values | From screening to hospitalization and follow up periods, assessed up to 43 days
  Changes and their clinical meaningfulness in clinical laboratory values: Hematology, Biochemistry, Urinalysis
Abnormal electrocardiogram (ECG) readings and their clinical meaningfulness | From screening to hospitalization and follow up periods, assessed up to 43 days
  ECG intervals (PR [PQ], QRS, QT, QTcF) and heart rate
Changes of ECG parameters and their clinical meaningfulness | From screening to hospitalization and follow up periods, assessed up to 43 days
  ECG intervals (PR [PQ], QRS, QT, QTcF), heart rate, T-wave morphology and U-wave morphology.
Abnormal vital signs and their clinical meaningfulness | From screening to hospitalization and follow up periods, assessed up to 43 days
  Blood pressure, heart rate and body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Sam Francis, Doctor, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia